CLINICAL TRIAL: NCT05375292
Title: Efficacy of Pre-Operative Prehabilitation in Patients Undergoing Open Surgery for Abdominal Aortic Aneurysm
Brief Title: Evaluation of the Impact of Prehabilitation on Recovery Following Open Surgery for Abdominal Aortic Aneurysm
Acronym: EPOP-AORTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/21/0618
Record Dates: First submitted 2022-05-05; First posted 2022-05-16 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: aaa; prehabilitation; quality of life; physical therapy; open surgery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Alzheimer Disease | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Monocentric, interventional, randomized, controlled, open study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREHABILITATION GROUP (Experimental): Initial visit with the adaptive rehabilitation physician, 6-8 weeks prior to surgery:
  * Clinical examination with Wood classification description of impairments, activity limits and participation restrictions.
  * Assessment of environmental resources
  * Definition with the patient of the extended ambulatory pre-habilitation protocol, identification with the post-operative rehabilitation pathway,
  * Provide the patient with a follow-up workbook of the personalized pre-approval protocol and, if the patient's condition requires it, orders for physiotherapy.
  Then apply the ambulatory pre-approval protocol defined with the adaptive rehabilitation physician.
  - Post-operative follow-up visits with the surgeon (gathering the necessary information for comparative follow-up).
  Mail-out of WHODAS 2.0 EQ-5D-5L and DIJON questionnaires at 3 and 6 months post-operative.
  Interventions: Other: PREHABILITATION
- CONTROL GROUP (No Intervention): Support without pre-approval with application of other common practices of the service.
  Post-operative follow-up visits with the surgeon (gathering the necessary information for comparative follow-up).
  Mail-out of WHODAS 2.0 EQ-5D-5L and DIJON questionnaires at 3 and 6 months post-operative.

INTERVENTIONS:
Other: PREHABILITATION — Customized program made by the physical therapist based on the first visit.
  It includes 3 parts :
  1. Nutrition advices that ensures adequate caloric and protein intake to support muscle anabolism
  2. Muscle building over a few sessions with a physiotherapist to learn exercises and then independently redo them
  3. Cardio-respiratory endurance exercises.
  Arms: PREHABILITATION GROUP

SUMMARY:
This is a pilot, prospective, randomized control trial that aim to provide a first estimation of the 3-month post-operative variation in the functional recovery of patients who benefited from an outpatient pre-habilitation program and patients who did not benefit from it.

DETAILED DESCRIPTION:
Open surgery of abdominal aortic aneurysms (AAA) is the reference treatment in a large number of cases. This is a heavy procedure performed in patients around 70 years of age.

In post-operative open aortic surgery, a stay in aftercare and rehabilitation is often necessary, especially in fragile patients.

The goal is to increase the patient's overall functional status to allow him to move away from the threshold below which he loses his independence for activities of daily living.

The pre-habilitation protocol includes 3 parts :

1. Oral nutrition ensures adequate caloric and protein intake to support muscle anabolism
2. Muscle building over a few sessions with a liberal physiotherapist to learn exercises and then independently
3. Cardio-respiratory endurance.

For the experimental group:

Initial visit with adaptive rehabilitation physician, 6-8 weeks prior to surgery:

* Clinical examination with Wood classification - limits and restrictions.
* Assessment of environmental resources
* Definition pre-habilitation protocol and post-operative rehabilitation pathway
* application of the ambulatory pre-approval protocol defined with the adaptive rehabilitation physician.

For the control group:

Support without pre-approval with application of other common practices of the service.

Follow up of both groups:

Post-operative follow-up visits with the surgeon (gathering the necessary information for comparative follow-up).

Mail-out of World Health Organisation Disability Assessment Schedule (WHODAS) 2.0, Euro Qol (EQ)-5D-5L and DIJON questionnaires at 3 and 6 months post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an abdominal aortic aneurysm (Thoraco-abdominal aneurysm type 4/Supra renal/Juxta-renal/Sub renal) treated with conventional surgery.
* Surgical indication of aneurysm by size (50-55mm)

Exclusion Criteria:

- Patient requiring urgent management that does not allow for a pre-authorisation protocol of at least 6 weeks.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
functional WHODAS 2.0 score | T0 : Right after the open surgery for AAA
  the WHODAS 2.0 score ranges from 12 to 60 : 12 representing no difficulty at all, 60 representing worst difficulty to engage in usual activities
functional WHODAS 2.0 score | 3 months after the open surgery for AAA
  the WHODAS 2.0 score ranges from 12 to 60 : 12 representing no difficulty at all, 60 representing worst difficulty to engage in usual activities

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Hostalrich, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Uh Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No